CLINICAL TRIAL: NCT02098122
Title: Upper Limb Activity in Human SCI Rehabilitation
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Foundation Wings For Life (Other); IRP International Foundation for Research in Paraplegia (Unknown)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-2013-0202/PB2016-00338
Record Dates: First submitted 2014-03-13; First posted 2014-03-27 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Tetraplegia
- Paraplegia

SUMMARY:
Functional recovery following SCI in adults is limited. Improvements in the quality of life of affected persons are associated with the recovery of functions that allow independent living, for example use of the arms and hands. Rehabilitative training has been shown to aid upper limb recovery. However, there are likely vast differences in the amount of time individuals spend actively training (during rehabilitation sessions in the clinic) and what they do in their non-training time (during daily life). The activity, or lack of, during the non-training period could interfere (positively or negatively), with the specific training in the rehabilitation session. However, there is little information available about this.

Inertial measurement units are increasingly being used in human movement and rehabilitation research. The use of such technology is a promising approach to rapidly and discreetly collect objective movement information. The investigators plan to introduce a novel, long-term, activity sensor into clinical SCI rehabilitation. The investigators use this sensor to precisely measure movement of the upper limb over extended periods of time. Upper limb activity recordings from these sensors allow us to detail the amount and duration of activity during specific periods of upper limb rehabilitation and recovery.

The investigators aim is to measure upper limb activity. The investigators aim to track changes in the activity of the upper limb during recovery and rehabilitation in patients with cervical SCI as well as collect reference values of upper limb activity in chronic sufferers. The recordings from this activity sensor will provide a more detailed understanding of how everyday upper limb activity contributes to functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Tetraplegic and paraplegic subjects.
* Males and females aged 18 or older.
* Acute (defined here as <90 days after admission of SCI) for the longitudinal follow-up study, as well as chronic (defined here as >90 days after admission of SCI) for the cross-sectional study, all levels of injury, complete and incomplete, traumatic and non-traumatic injuries.
* Good enough cognitive ability to be able to follow simple verbal instructions.
* Signed informed consent before study onset.

Exclusion Criteria:

* A neurological disease other than SCI, which is expected to affect the upper limb function, i.e. plexus paresis.
* An orthopaedic or rheumatologic disease, e.g. osteoarthritis, which is expected to affect the upper limb function.
* Pre-morbid on-going major depression or psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spinal Cord Injured Subjects
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Change of physical activity levels | Cross-sectional and longitudinal (2weeks, 1month, 3months, 6months, 12months)
  Changes of activity levels will be assessed by calculating activity counts from the accelerometer data.

CONTACTS AND LOCATIONS:
Overall Officials: Armin Curt, MD, Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Brogioli M, Schneider S, Popp WL, Albisser U, Brust AK, Velstra IM, Gassert R, Curt A, Starkey ML. Monitoring Upper Limb Recovery after Cervical Spinal Cord Injury: Insights beyond Assessment Scores. Front Neurol. 2016 Aug 31;7:142. doi: 10.3389/fneur.2016.00142. eCollection 2016. PMID 27630612
- [Background] Brogioli M, Popp WL, Schneider S, Albisser U, Brust AK, Frotzler A, Gassert R, Curt A, Starkey ML. Multi-Day Recordings of Wearable Sensors Are Valid and Sensitive Measures of Function and Independence in Human Spinal Cord Injury. J Neurotrauma. 2017 Mar 15;34(6):1141-1148. doi: 10.1089/neu.2016.4583. Epub 2016 Oct 12. PMID 27533063
- [Background] Brogioli M, Popp WL, Albisser U, Brust AK, Frotzler A, Gassert R, Curt A, Starkey ML. Novel Sensor Technology To Assess Independence and Limb-Use Laterality in Cervical Spinal Cord Injury. J Neurotrauma. 2016 Nov 1;33(21):1950-1957. doi: 10.1089/neu.2015.4362. Epub 2016 May 16. PMID 27025797
- [Background] Popp WL, Brogioli M, Leuenberger K, Albisser U, Frotzler A, Curt A, Gassert R, Starkey ML. A novel algorithm for detecting active propulsion in wheelchair users following spinal cord injury. Med Eng Phys. 2016 Mar;38(3):267-74. doi: 10.1016/j.medengphy.2015.12.011. Epub 2016 Feb 8. PMID 26868046